CLINICAL TRIAL: NCT06486311
Title: Assessment of Stability Using Satellite Implant for Immediate Loading in Posterior Mandible
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Tallah Selim Labib Kaream, dentist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: satellite implant
Record Dates: First submitted 2024-06-22; First posted 2024-07-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Novel Implant for Immediate Load in Posterior Mandible
Keywords: "Micro fixation "; "Immediate Loading"; "Posterior Mandible"; "Stability"

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment stability of satellite implant (Experimental): Satellite implant is connecting microplate is attached to the implant's supra structure placed on the adjacent alveolus. Miniature "satellite" implant screws are inserted at approximal cortical sites to give the implant additional stability
  Interventions: Procedure: satellite implant

INTERVENTIONS:
Procedure: satellite implant — Satellite implant is a additional holding component as a stabilizer to provide a polygonal support to distribute forces and moments on single-standing implants give the implant sufficient resistance to withstand masticatory forces or at least keep it in a stable position during an unloaded healing period to achieve stabilization and subsequent osseointegration of implants.

SUMMARY:
The research aims to evaluate the long-term effectiveness of satellite implants in the posterior mandible by assessing the levels of crestal bone after six months of first loading and secondary stability issues at fourth-month , primary stability at time of implant loading . In particular, the primary outcome of this study is to assessment stability of satellite implants, which will be evaluated by anycheck device.

DETAILED DESCRIPTION:
satellite dental implants show potential for improving stability, and reducing crestal bone loss in the posterior mandible site, it offers effective solution for cases where primary stability is compromised due to poor bone quality or quantity. By providing additional support and anchorage, they enhance the overall stability of the implant, reducing the risk of failure and allowing for successful immediate loading. clinical evidence for their efficacy is still lacking. This prospective case series intends to fill this gap by evaluating crestal bone levels and stability factors in patients who are getting satellite implants for immediate loading in the posterior mandible. The results will improve clinical recommendations and practice for implant placements in the posterior mandible.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implants for the posterior mandible.
* Patients aged between 18-45 years old.
* Implants must be at least 8mm in length.
* A sufficient quantity and distribution of implants to enable cross-arch stability.
* Implants must have good initial stability, with insertion torques ranging from 35 to 50 N/cm.
* Sufficient bone for implant placement and plate fixation.
* Patient able to give informed consent.
* Sufficient inter-arch space.

Exclusion Criteria:

* Contraindications to implant surgery in general.
* Bruxism.
* Immunosuppression.
* History of radiation to the head and neck region.
* Uncontrolled diabetes.
* Heavy smokers (more than ten cigarettes per day).
* Poor oral hygiene.
* Current or previous bisphosphonate therapy.
* Substance abuse.
* Mental illness.
* Failure to complete 6-month follow-up.
* Pregnancy or breastfeeding.
* Insertion torque of less than 35 N/cm.
* Removal of interim repair during the osseointegration stage.
* Patients suffering from parafunctional behaviors.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-22 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Stability Using Satellite Implant for Immediate Loading in Posterior Mandible | Immediately post-implantation
  After the insertion of the satellite implant, primary stability will be assessed at the time of implant loading using the "AnyCheck" device (Neo Biotech, Seoul, Korea). Introduced in 2017, the AnyCheck device evaluates implant stability through a damping capacity assessment method. It functions by striking the healing abutment six times over a span of three seconds. The contact duration between the impacting rod and the healing abutment is measured and converted into Implant Stability Test (IST) values. These values are quantified on a scale from 1 to 99, where higher IST values indicate greater implant stability or lower mobility. This quantitative measure provides a precise, reproducible method to assess the outcome of implant stability immediately after placement.

SECONDARY OUTCOMES:
Assessment of Stability Using Satellite Implant for Immediate Loading in Posterior Mandible | The secondary stability is assessed four months post-implantation for each patient.
  Assessment Tool: Secondary stability will be assessed using the "AnyCheck" device (Neo Biotech, Seoul, Korea). Introduced in 2017, this device specifically measures the damping capacity to evaluate implant stability.
  Method: After the removal of the satellite implant four months post-procedure, the AnyCheck device will be employed to measure the secondary stability. The device operates by striking the healing abutment six times over a three-second period. The duration of contact between the impacting rod and the healing abutment is recorded.
  Measurement Scale: The recorded contact time is then converted into Implant Stability Test (IST) values, which are displayed on a scale from 1 to 99. Higher IST values indicate greater implant stability, reflecting lower mobility of the implant within the bone.

OTHER OUTCOMES:
Assessment of Stability Using Satellite Implant for Immediate Loading in Posterior Mandible | Crestal bone loss will be assessed at baseline (immediately post-implantation) and six months after the implant procedure. This timeframe allows for the monitoring of early bone remodeling and loss around the satellite implant.
  Measurement Tool: CBCT combined with calibrated dental software.
  Method: Crestal bone level will be precisely measured by assessing the interproximal height of bone. This is defined as the distance between the apical end of the first thread of the implant and the most coronal point of the interproximal crestal bone, both buccally and lingually. Measurements will be taken using digital periapical radiographs, which provide high-resolution images allowing for accurate assessment of bone levels.
  Data Analysis: The height of the crestal bone will be recorded in millimeters. For each implant, the mean of the buccal and lingual bone heights will be calculated to determine the average crestal bone loss.
  Measurement Scale: Measurements will be recorded in millimeters to provide a precise quantitative assessment of bone loss.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.hesham shalakamy, lecturer, Principal Investigator — • Lecturer of Oral and Maxillofacial Surgery- Cairo University
Locations (1):
- Aya Tallah Selim Labib Kaream, Cairo, Shrouk, Egypt

REFERENCES:
- [Background] Engelke W, Stahr S, Schwarzwaller W. Enhancement of primary stability of dental implants using cortical satellite implants. Implant Dent. 2002;11(1):52-7. doi: 10.1097/00008505-200201000-00014. PMID 11915545
- [Background] Engelke W, Decco OA, de las Mercedes Capobianco M, Schwarzwaller W, Villavicencio MM. Immediate occlusal loading of freestanding implants using cortical satellite implants: preliminary report of a prospective study. Implant Dent. 2005 Mar;14(1):50-7. doi: 10.1097/01.id.0000154796.97355.2d. PMID 15764945